CLINICAL TRIAL: NCT00053300
Title: Phase II Trial of Daily Thalidomide in Extensive Stage Small Cell Lung Cancer Patients Achieving a Complete or Partial Response to Induction Chemotherapy
Brief Title: Thalidomide in Treating Patients With Extensive-Stage Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Afshin Dowlati, MD, Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CWRU1502; P30CA043703 (NIH); CASE-CWRU-1502 (Other: Case Comprehensive Cancer Center); CELGENE-CWRU-1502; CASE-1502 (Other: Case Comprehensive Cancer Center)
Record Dates: First submitted 2003-01-27; First posted 2003-01-28 (Estimated); Last update posted 2010-06-10 (Estimated); Status verified 2010-06

CONDITIONS: Lung Cancer
Keywords: extensive stage small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Thalidomide; Chemotherapy, Adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: thalidomide — oral thalidomide daily beginning 3-4 weeks after completion of induction chemotherapy. Treatment continues for 1 year in the absence of disease progression or unacceptable toxicity
Procedure: adjuvant therapy — Patients receive oral thalidomide daily beginning 3-4 weeks after completion of induction chemotherapy. Treatment continues for 1 year in the absence of disease progression or unacceptable toxicity.

SUMMARY:
RATIONALE: Thalidomide may stop the growth of cancer by stopping blood flow to the tumor.

PURPOSE: Phase II trial to study the effectiveness of thalidomide in treating patients who have extensive-stage small cell lung cancer that has responded to previous chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the effect of thalidomide on time to disease progression and survival in patients with extensive-stage small cell lung cancer who achieve a complete or partial response to induction chemotherapy.
* Determine the toxicity of this drug in these patients.

OUTLINE: This is an open-label study.

Patients receive oral thalidomide daily beginning 3-4 weeks after completion of induction chemotherapy. Treatment continues for 1 year in the absence of disease progression or unacceptable toxicity

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study within approximately 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of extensive-stage small cell lung cancer
* Complete or partial response after 4-6 courses of induction chemotherapy

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* At least 2 months

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use 2 effective methods of contraception for at least 4 weeks before, during, and for at least 4 weeks after study
* No greater than grade 1 peripheral neuropathy

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2002-08; Primary Completion 2005-11 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Disease response | every 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Afshin Dowlati, MD, Study Chair — Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio

REFERENCES:
- [Result] Cooney MM, Subbiah S, Chapman R, et al.: Phase II trial of maintenance daily oral thalidomide in patients with extensive-stage small cell lung cancer (ES-SCLC) in remission. [Abstract] J Clin Oncol 23 (Suppl 16): A-7166, 661s, 2005.